CLINICAL TRIAL: NCT01419808
Title: Vascularized vs. Non-vascularized Bone Grafting in the Treatment of Proximal Pole Scaphoid Non Unions: A Prospective Randomized Trial
Brief Title: Vascularized Versus Non-Vascularized Bone Grafts in Treating Proximal Pole Scaphoid Non Unions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hand and Upper Limb Clinic, Canada (Network)
Responsible Party: Dr. Ruby Grewal, Hand and Upper limb Centre, St Joseph's Health Care
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HULCscaphoid
Record Dates: First submitted 2011-08-09; First posted 2011-08-18 (Estimated); Last update posted 2011-08-18 (Estimated); Status verified 2011-08

CONDITIONS: Scaphoid Non-Unions
Keywords: Scaphoid; Non-Union; Proximal pole; Bone Graft; Vascularized; Non-Vascularized; PREE
MeSH Terms: conditions — Neovascularization, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vascularized Bone Graft (Active Comparator): Patients randomized to a vascularized bone graft will undergo a 1, 2-ICRSA vascularized bone graft based upon the 1,2 supra-retinacular vessels as described by Zaidemberg . (9. Zaidemberg C, Siebert JW, Angrigiani C. A new vascularized bone graft for scaphoid nonunion. J Hand Surg. 1991; 16A: 474-478.)
  Interventions: Procedure: Vascularized Bone Graft
- Non-Vascularized Bone Graft (Active Comparator): Patients randomized to the non-vascularized group will undergo trapezoidal bone grafting from the iliac crest as described by Fernandez . (10. Fernandez DL. A technique for anterior wedge-shaped grafts for scaphoid nonunions with carpal instability. J Hand Surg [Am]. 1984 Sep;9(5):733-7.)
  Interventions: Procedure: Non-Vascularized Bone Graft

INTERVENTIONS:
Procedure: Vascularized Bone Graft — Vascularized bone graft in the treatment of Scaphoid Non-Union
  Arms: Vascularized Bone Graft
Procedure: Non-Vascularized Bone Graft — Non-Vascularized Bone Graft in the treatment of Scaphoid Non-unions
  Arms: Non-Vascularized Bone Graft

SUMMARY:
The purpose of this study is to investigate whether treatment of scaphoid non-unions with a vascularized bone grafts improves patient reported pain and disability compared to treatment with a non-vascularized bone graft. Secondary objectives are to examine if there is any difference in the overall rate and time to union, range of motion, grip strength, or complication rates between the two groups.

In addition, this is the first prospective randomized study to directly compare the two techniques. This is also the first study to use standardized methods of assessing union (based on computerized tomography), standardized methods of collecting objective patient data, and utilizing validated patient questionnaires to assess pain and disability.

ELIGIBILITY:
Inclusion Criteria:

* The primary inclusion criterion is any scaphoid waist or proximal pole non-union in a patient receiving a recommendation for operative treatment. Non-union is defined as <10% bony union across the fracture site on sagittal computerized tomography (CT) after at least 16 weeks of appropriate non-operative treatment or morphologic features on plain x-ray and CT (resorption and sclerosis at the fracture site, significant cyst formation) confirming non-union.

Exclusion Criteria:

* radiologic evidence of significant scaphoid non-union advanced collapse (SNAC) wrist arthritis
* fragmentation of the proximal pole

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-09; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Patient Rated Wrist Evaluation | Change in PRWE score at time of Surgery (day 1) compared to two years post operation.
  Patients will fill out the patient rated wrist Evaluation Questionnaire

SECONDARY OUTCOMES:
Objective Measures | Change in strength, ROM, and Dexterity from time of surgery (day 1) compared to two years post operation.
  * ROM
  * Grip Strength
  * Dexterity

CONTACTS AND LOCATIONS:
Overall Officials: Ruby Grewal, MD, FRCSC, Principal Investigator — Hand and Upper Limb Centre, St. Joseph's Health Care
Locations (1):
- Hand and Upper Limb Centre, St Joseph's Health Care, London, Ontario, Canada

REFERENCES:
- [Derived] Fan S, Suh N, MacDermid JC, Ross D, Grewal R. Vascularized versus non-vascularized bone grafting for scaphoid nonunion without avascular necrosis: a randomized clinical trial. J Hand Surg Eur Vol. 2023 Jul;48(7):648-653. doi: 10.1177/17531934231158992. Epub 2023 Mar 1. PMID 36861269